CLINICAL TRIAL: NCT04588831
Title: Comfort and Wearability of Custom-fitted, Mouth-formed and Pre-fabricated Mouthguards for Patients Undergoing Fixed Appliance Therapy: a Single-center, Single Blind Randomized Cross-over Trial
Brief Title: Comfort and Wearability of Custom-fitted, Mouth-formed and Pre-fabricated Mouthguards for Patients Undergoing Fixed Appliance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RoyalSurreyNHS
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Mouth Protectors
Keywords: mouth protectors
MeSH Terms: interventions — Mouth Protectors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-fabricated (Experimental)
  Interventions: Device: Mouthguard
- Mouth-formed (Experimental)
  Interventions: Device: Mouthguard
- Custom-fitted (Experimental)
  Interventions: Device: Mouthguard

INTERVENTIONS:
Device: Mouthguard — Protective device for orofacial complex for patients playing contact sports

SUMMARY:
There is no current evidence on the comfort or wearability of orthodontic mouthguards. These mouthguards adapt to the mouth without the need for dental impressions and laboratory facilities and are suggested to be more comfortable for orthodontic patients by allowing the teeth to move during treatment without the need for them to be replaced regularly during treatment. This study aims to assess and compare the comfort and wearability of orthodontic mouthguards with custom-fitted mouthguards. The results of this study will allow orthodontists to provide evidence-based information to individuals undergoing fixed appliance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing active orthodontic treatment with pre-adjusted edgewise fixed appliances only for a minimum period of 9 months
* Playing sports where the use of a mouthguard is recommended
* Playing at least 120 minutes of sport (match or training) during a 6-8 week period
* Class I, II or mild III (edge-to-edge) incisor malocclusion
* Able to complete a VAS questionnaire
* No diagnosed sensory processing disorder

Exclusion Criteria:

* Undergoing active orthodontic treatment that is not pre-adjusted edgewise fixed appliances, or requires a fixed expander, or treatment is likely to be completed within 9 months
* Playing sports where the use of a mouthguard is not recommended Playing less than 120 minutes of sport (match or training) during a 6-8 week period
* Moderate to severe class III (reverse overjet) incisor malocclusion
* Unable to complete a VAS questionnaire
* Have a diagnosed sensory processing disorder

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Comfort and wearability of all three mouthguards | 4 years
  The primary and only outcome of this study was the response to each question of the administered questionnaire.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kalra A, Harrington C, Minhas G, Papageorgiou SN, Cobourne MT. Wearability and preference of mouthguard during sport in patients undergoing orthodontic treatment with fixed appliances: a randomized clinical trial. Eur J Orthod. 2022 Jan 25;44(1):101-109. doi: 10.1093/ejo/cjab062. PMID 34748017